CLINICAL TRIAL: NCT02735460
Title: Single-center Usability Study of the Overground Gait and Balance Training Device Andago V2.0 in Patients With Gait Disorder After Stroke at a Center for Neurological Rehabilitation
Brief Title: Usability of Andago V2.0 in Gait Rehabilitation of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehaklinik Zihlschlacht AG (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RZI_01_2015
Record Dates: First submitted 2016-03-15; First posted 2016-04-12 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Brain Ischemia; Intracranial Haemorrhage
MeSH Terms: conditions — Brain Ischemia; Intracranial Hemorrhages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Experimental): In this arm the Andago V2.0 is used.
  Interventions: Device: Andago V2.0

INTERVENTIONS:
Device: Andago V2.0 — The Andago V2.0 is tested in 2 sessions, the first being a training session to define the probably optimal settings for the subsequent therapy session. In the therapy session the participant performs a specific parcours. Usually this parcours can be done within 10 minutes. However, the session is stopped as soon as the patient feels too exhausted or becomes too weary.

SUMMARY:
Andago V2.0 is a recently developed overground gait and balance training device. Many patients in neurorehabilitation suffer from gait disorders, most typically after stroke. Since pharmacological therapies are basically not available, neurorehabilitation plays an important role in the treatment of such patients. The Andago V2.0 may represent a useful device in the rehabilitation of stroke and other neurological patients featuring a severe gait disorder. Therefore a study has been designed to investigate the usability of the Andago V2.0 in the setting of a neurorehabilitation clinic. The primary outcomes of this study are the usability and acceptance of the investigational medical device (IMD). Usability is mainly measured by the time spent for the set-up and release of the participant, achieved training times and distances, the number of stumbles, collisions and emergency stops and the error messages during the session. Besides patient and therapist satisfaction with the Andago V2.0 is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Primary diagnosis of cerebral infarction (ICD-10: I63.0-I63.9) or intracerebral haemorrhage (ICD-10: I61.0-I69.9) independent of its location, age or cause
* Gait disorder defined by a category of 1 to 3 on the Functional Ambulation Classification (FAC) (17)
* Age above 18 years
* Admission to Rehaklinik Zihlschlacht for in-patient neurorehabilitation

Exclusion Criteria:

* Inability of the participant to understand the informed consent or to follow the procedures of the study, e.g., due to language problems, psychiatric disorders, cognitive impairment or aphasia (item 9 of the National Institute of Health Stroke Scale (NIHSS) ≥2)
* Weight >135 kg
* Height >200 cm
* Bone fragility (e.g., non-consolidated fractures or osteotomies including craniotomies, osteopenia, osteoporosis or symptoms or indices in the patient history that infer a higher risk of bone density reduction)
* Unstable arthroplasty
* Uncontrolled knee or ankle instability that would still pose a danger despite the Body Weight Support (BWS) (especially lateral instability)
* Lack of head control
* Joint contractures
* Relevant differences in leg length
* Skin lesions (including pressure sores or enteric stomata) in areas of contact with harness support or lower extremity loading (feet)
* Relevant sensory impairment in the lower limbs and trunk, especially with reduced pain sensation
* Recent history or significant risk of seizures
* Relevant cardiovascular conditions, e.g., cardiac insufficiency and thoracotomy, uncontrolled orthostatic hypotension or other circulatory problems, vascular disorders of the lower limbs
* Mechanical ventilation
* Long-term infusions (e.g., baclofen pump, other intrathecal pumps)
* Any medical condition preventing active rehabilitation and/or the use of the Andago V2.0 (e.g., respiratory disease, pregnancy, orthopedic conditions, infections or inflammatory disorders, osteomyelitis)
* Participation in another interventional study within the 30 days preceding and during the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
Usability of the IMD according to the number of participants that are able to use the Andago V2.0 | 3 weeks
Acceptance of the IMD as measured by a therapist satisfaction questionnaire | 3 weeks
Acceptance of the IMD as measured by a patient satisfaction questionnaire | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Marks, Principal Investigator — Rehaklinik Zihlschlacht
Locations (1):
- Rehaklinik Zihlschlacht, Center for Neurological Rehabilitation, Zihlschlacht, Switzerland

IPD SHARING:
Plan to Share IPD: No